CLINICAL TRIAL: NCT04660825
Title: The Efficacy of a Resistance Band Exercise Intervention to Improve Vertebral Fracture Risk Facts in Post-menopausal Women
Brief Title: Development and Evaluation of an Exercise Intervention for Prevention of Vertebral Osteoporosis and Deformity in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Katherine Brooke-Wavell, Senior Lecturer in Human Biology, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R18-P094
Record Dates: First submitted 2020-06-09; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Osteoporosis; Osteoporotic Fracture of Vertebra; Postural, Thoracic Kyphosis
Keywords: Resistance band exercise; High intensity; Osteoporosis; DXA; Bone; Exercise
MeSH Terms: conditions — Osteoporosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study will be a randomised controlled trial of a six-month exercise intervention. Following screening and baseline measurements, participants will be randomly assigned to exercise or control groups, allocated in 2:1 ratio. Randomisation will conducted using computer algorithm. The exercise group will be requested to complete the intervention as detailed below whilst the control group maintain their usual lifestyle.
  Participants will complete a six-month programme of muscle-strengthening exercises using resistance bands. Exercises will be introduced through group sessions run three times per week, some of which could be substituted by home exercise supported by an exercise booklet and video.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity resistance band exercise (Experimental): Randomly assigned as exercise group, exercise intervention. This will be a progressive exercise programme with the aim being to participate three times per week, one in a group session and two in-home sessions.
  Interventions: Other: A resistance band exercise programme
- Non resistance band exercise (Experimental): Randomly assigned non-exercise group
  Interventions: Other: Control

INTERVENTIONS:
Other: A resistance band exercise programme — A resistance band based exercise programme lasting six months
  Arms: High intensity resistance band exercise
Other: Control — Maintained usual physical activity
  Arms: Non resistance band exercise

SUMMARY:
Osteoporotic fractures of the vertebrae (bones in the back) cause substantial pain and disability. Exercise could help to prevent these fractures by increasing bone strength and improving posture. Unfortunately, not all exercises strengthen bone. Exercises that do work (e.g. heavy weight lifting) are not popular with women at risk of osteoporosis. The investigators will develop a feasible exercise programme that can be done at a community centre or at home, using resistance bands. The investigators will involve women in designing the programme and incorporate strategies to support behaviour change. The investigators will then examine whether the programme improves bone density, posture or muscle strength in eighty women. Half the women, chosen at random, will take up exercise whilst the remaining half act as a control group. The investigators will take bone scans to determine bone density, and measure spinal curvature and strength, before and after the six- month programme. Findings will be useful in making recommendations as to which types of exercise increase spine bone density and will help to design future research on maximising vertebral strength. If significant benefits are seen, the investigators will develop resources such as booklets and videos so that the intervention can be widely available.

DETAILED DESCRIPTION:
Healthy, post-menopausal elderly women without other conditions restricting them from completing an exercise intervention. Inclusion criteria will be: Aged 60-80 and postmenopausal for at least 5 years, not taking/eligible for osteoporosis medication. Exclusion criteria will be: regular (>once per week) participation in high impact or high load resistance training, any disease or medication that contraindicates exercise or affects bone metabolism, meet UK criteria for pharmaceutical treatment of osteoporosis (will be referred to GP for treatment). The primary outcome measure will be AP lumbar spine (L1-4) BMD, measured by DXA using a GE Lunar iDXA densitometer. Secondary outcomes will include: BMD at femoral neck and lateral BMD of vertebra and hip structural parameters by DXA. Vertebral morphometry and dimensions, and total and regional body composition (bone, fat and lean masses), spinal curvature will be assessed from lateral DXA scans using statistical shape modelling (SSM) and the Cobb angle will be calculated as a measure of kyphosis, previous and current bone relevant physical activity will be assessed using a validated questionnaire, physical performance will be assessed using the Short Physical Performance Battery and functional mobility will be assessed using the Senior Fitness Test (SFT), peak force developed during exercises will be assessed by performing exercise using a resistance band of the current weight instrumented using a spring balance, postural sway will be assessed by measuring the movement of the centre of mass (COM), centre of foot pressure (COP), body segment through force platforms.

The intervention group will be asked to take up a six-month programme of muscle strengthening exercises using resistance bands. Exercises will be introduced through group sessions run three times per week, some of which could be substituted by home exercise supported by an exercise booklet and video. The intervention will consist of initial spinal extension and core strengthening exercises to ensure good posture and form (e.g. thoracic spine extension and abdominal exercise avoiding spinal flexion). Exercises that increased BMD will be adapted for resistance bands, initially at low intensity to allow development of good technique. Intensity will be increased gradually by employing bands of greater stiffness until participants can only complete 8 repetitions without a break. Once participants can attain 12 repetitions, intensity will be progressed by using a higher strength band. Participants will be advised in technique and progression at group sessions, to support transition to independent exercise by the end of the study.

The intervention will include a behaviour change component that considers capability, opportunity and motivation using the Behaviour Change Wheel framework by using the taxonomy of behaviour change interventions to identify the most appropriate strategies for facilitating behaviour change. The nature of the intervention considers the social and physical limitations to opportunity to exercise, and physical and psychological capability as identified in the qualitative phase by incorporating a group component to exercise and avoiding settings such as a gym. To accord with the practical and environmental factors identified, sessions will be offered at a variety of times of day. Explanations of safety of exercise with low BMD and purpose of the exercises in the group class and booklet/video will underpin knowledge aspects. Participants will be encouraged to be involved in goal setting and action planning. This will be supported using text reminders and motivational messages or other support strategies. Feedback in group sessions will also reinforce reflective motivation. Support and implementation strategies will be continuously reviewed based upon findings in initial participants. The control group will be asked to continue their usual exercise and dietary habits as if they were not participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-80 and postmenopausal for at least 5 years
* Not taking/eligible for osteoporosis medication

Exclusion Criteria:

* Regular (>once per week) participation in high impact or high load resistance training.
* Any disease or medication or injury that contraindicates exercise or affects bone metabolism.
* Meet UK criteria for pharmaceutical treatment of osteoporosis (will be referred to GP for treatment).

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in AP lumbar spine (L1-4) bone mineral density (g/cm2) | Baseline measurement and 6 month follow-up measurements
  Lumbar spine bone mineral density measured by DXA using a GE Lunar iDXA densitometer

SECONDARY OUTCOMES:
Change in AP lumbar spine bone mineral density (g/cm2) | Baseline measurement and 6 month follow-up measurements
  DXA scan: Measurement of lumbar spine bone mineral density (g/cm2)
Change in AP lumbar spine mineral content (g) | Baseline measurement and 6 month follow-up measurements
  DXA scan: Measurement of lumbar spine mineral content (g)
Change in femoral neck bone mineral density (g/cm2) | Baseline measurement and 6 month follow-up measurements
  DXA scan: Measurement of femoral neck bone mineral density (g/cm2)
Change in femoral neck bone mineral content (g) | Baseline measurement and 6 month follow-up measurements
  DXA scan: Measurement of femoral neck bone mineral content (g)
Change in spinal curvature (°) | Baseline measurement, 3 months and 6 month follow-up measurements
  Spinal curvature will be assessed from lateral DXA scans using the Cobb angle as a measure of kyphosis.
Change in chair stand (sec) | Baseline measurement, 3 months and 6 months follow-up measurements
  Chair stand: Time taken to stand up and sit down as quickly as possible 5 times.
Change in gait speed (sec) | Baseline measurement, 3 months and 6 months follow-up measurements
  Timed walk (Gait speed): Time taken to walk 8-feet (2.44metres)
Change in balance (sec) | Baseline measurement, 3 months and 6 months follow-up measurements
  Tandem balance: Ability to balance unsupported for 10 seconds with feet in three different positions (i.e side by side stands [feet together], semi tandem and full tandem).
Change in timed up and go (sec) | Baseline measurement, 3 months and 6 months follow-up measurements
  Timed up and go: Time taken to rise from a chair, walk three metres away, turn and walk back to the chair and sit down again.
Change in back scratch (cm) | Baseline measurement, 3 months and 6 months follow-up measurements
  Back scratch: Distance between hands when reaching both arms behind the back: one arm upwards, one down.
Change in arm curls (rep) | Baseline measurement, 3 months and 6 months follow-up measurements
  Arm curls: Number of bicep curls that can be completed in 30s with a 2.25kg dumbbell.
Change in Posture sway (mm) | Baseline measurement, 3 months and 6 months follow-up measurements
  Postural sway will be assessed by measuring the movement of the centre of foot pressure (COP) using a force platform. Measurements will be repeated 30 seconds in four conditions: eyes open, firm surface eyes closed, firm surface eyes open, compliant surface eyes closed, compliant surface.
Change in Trunk extensor strength (N) | Baseline measurement, 3 months and 6 months follow-up measurements
  Trunk extensor strength will be using a handheld dynamometer. Participant will be asked to lie prone on a couch and push upward against the dynamometer which is mounted on a custom built frame. Participants will be allowed three attempts and the maximum force recorded.
Change in Trunk extensor endurance (sec) | Baseline measurement, 3 months and 6 months follow-up measurements
  Back endurance in trunk extension will be assess with the participant lying prone. Participants will be asked to lift the upper body off the surface and hold for as long as possible. The time will be recorded.
Change in peak force (kg) | Baseline measurement, 3 months and 6 months follow-up measurements
  Peak force developed during exercises will be assessed by performing exercise using a resistance band of the current weight instrumented using a spring balance.
A health screening questionnaire | Baseline measurement
  A health screening questionnaire will be used to assess suitability for the study
A PAR-Q questionnaire | Baseline measurement, 3 months and 6 months follow-up measurements
  A PAR-Q questionnaire will be used to check readiness to exercise
A CaQ Calcium intake questionnaire | Baseline measurement, 3 months and 6 months follow-up measurements
  A CaQ Calcium intake questionnaire will be used to estimate dietary calcium

CONTACTS AND LOCATIONS:
Locations (1):
- Donghyeon Seo, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No